CLINICAL TRIAL: NCT03807908
Title: The Short-term Effects of Taping During Pregnancy-related Low Back Pain, Pelvic Girdle Pain or Combined Pain
Brief Title: Effects of Taping on Pregnancy-related Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Carol Ann Weis, Researcher, Canadian Memorial Chiropractic College
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 182028
Record Dates: First submitted 2019-01-12; First posted 2019-01-17 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy; Low Back Pain; Pelvic Girdle Pain
Keywords: Pregnancy; Low back pain; Pelvic girdle pain; Kinesiotape
MeSH Terms: conditions — Low Back Pain; Pelvic Girdle Pain | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: The study will be a randomized clinical trial. As none of the current research delineates the 3 pains during pregnancy, it would be beneficial to further investigate the use of tape for LBP, PGP or combined pain during pregnancy. As such, the participants will be stratified upon pain presentation (via history and physical exam) and then randomized into either a treatment or sham protocol.
Who Masked: Participant
Masking Description: Once consent has been obtained the senior chiropractors will review the intake questionnaire with the patients, ask any pertinent questions they may have regarding the patient's personal medical history and current pain pattern and perform a physical exam to differentiate pain patterns for each participant.
  Following completion of baseline assessment and consent, participants will be stratified by their type of pain presentation and then be randomly allocated to 1 of the 2 intervention arms. Central randomization will be performed using stratified block randomization by the study biostatistician (SHJ) using SAS software*. To ensure that the allocation sequence is concealed from the researchers varying block sizes of 2, 4 and 6 will be used and the biostatistician will provide the trial coordinator with 3 series (1 for each stratum) of sequentially numbered sealed opaque envelopes containing the intervention allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Tape (Experimental): The intervention includes 3 strips of tape; 2 (1 on each side) placed vertically along the lumbar erectors and 1 horizontally at the posterior superior iliac spine.
  Subjects will wear the tape for as long as possible up to 5-7 days.
  Interventions: Other: Tape
- Sham Tape (Sham Comparator): One strip of tape will be applied horizontally to the thoracolumbar junction.
  Subjects will wear the tape for as long as possible up to 5-7 days.
  Interventions: Other: Sham Tape

INTERVENTIONS:
Other: Tape — The patient will be placed into maximal flexion of the lumbar spine prior to the tape being applied. The vertical strips will be applied on either side of spine, on the erector muscle group; from the lower PSIS with and end around the twelfth rib. The third strip of tape will be applied horizontally to superior to the posterior superior iliac spines (PSIS) and extend over the 2 vertical strips of tape. The tape will be gently rubbed to activate the adhesive.
  Five to 7 days later, one of the investigators will follow up with the subjects over the phone and administer a questionnaire that will assess their experience with the tape as well as the outcome measures (numeric rating scale and Oswestry Disability Index).
  Other Names: Kinesiotape
  Arms: Intervention Tape
Other: Sham Tape — One strip of tape will be applied horizontally to the thoracolumbar junction (at the level of the lower rib cage over the T12-L1 spinous processes) with no tape-tension. The tape will be gently rubbed to activate the adhesive.
  Five to 7 days later, one of the investigators will follow up with the subjects over the phone and administer a questionnaire that will assess their experience with the tape as well as the outcome measures (numeric rating scale and Oswestry Disability Index).
  Other Names: Kinesiotape
  Arms: Sham Tape

SUMMARY:
Back pain during pregnancy is common with up to 90% of pregnant women experiencing either low back pain (PLBP), pelvic girdle pain (PGP) or a combination of both pains. Although pregnant women seek out various forms of pain relief methods such as pain medication, exercise, education, pelvic support belts, and chiropractic treatments, there is limited evidence with regards to the efficacy of these treatments. Recently manual therapists, such as chiropractors, have used tape in an effort to relieve pain from musculoskeletal injuries with varying results. In the pregnant population, there have been limited studies to date on the role of taping and pregnancy-related back pain and none of this research delineates the efficacy of tape with respect to the 3 pain patterns experienced by pregnant women.

DETAILED DESCRIPTION:
This study is a randomized control trial with 3 main parts associated. 1) Initial visit: Potential participants will be recruited from 2 antenatal clinics at the participating hospital. A person from the circle of care will ask if they are interested in participating in a study regarding pregnancy-related LBP. Participants are pre-screened by a research investigator, If patients meet the eligibility criteria, they will be invited to participate. Research personnel will explain the study in full including the rationale (per the Project Consent Form), visit requirement, treatment protocol and follow-up. Once consent is obtained, a Pre-Visit Questionnaire will be administered while they are awaiting their antenatal appointment. 2) Physical exam and treatment: Following their appointment, research personnel will walk the participant to the Obstetrical Day Unit where the chiropractor will review the consent and questionnaire, perform a brief physical exam to ensure proper stratification of pain, randomized the participant (as pre-determined by the biostatistician) and apply the appropriate taping protocol (intervention vs sham). 3) Follow-up: Five to 7 days later, research personnel will follow-up with the participant by phone and administer a questionnaire pertaining to their experience with the taping protocol. The total visit should take no more than 30 minute

ELIGIBILITY:
Inclusion Criteria:

* Healthy females of childbearing age
* Currently experiencing a healthy, singleton pregnancy and are at 28 weeks of gestation or later
* Proficient competency in the English language

Exclusion Criteria:

* Does not wish to participate
* Carrying multiples
* Inability to understand the questionnaire due to a lack of understanding of the English language
* Allergy to tape and/or adhesives (acrylic copolymer)
* Prior spinal surgery
* A known and current disc pathology

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be experiencing a healthy, non-complicated pregnancy
Enrollment: 96 (Estimated)
Dates: Start 2019-07-31 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Numeric Pain Scale (Pain) to Numeric Pain Scale (Pain) 5-7 days later | 7 days
  Intensity of pain on a 0-10 scale; 0=no pain; 10=most severe pain
Change from baseline Oswestry Back Disability Index (ODI) to ODI 5-7 days later | 7 days
  Measure of a patient's functional disability

CONTACTS AND LOCATIONS:
Overall Officials: Carol Ann Weis, MSc, DC, Principal Investigator — Canadian Memorial Chiropractic College

IPD SHARING:
Plan to Share IPD: No